CLINICAL TRIAL: NCT07232875
Title: a Randomized, Controlled, Double-Blind, Multicenter Phase III Clinical Trial of HRS-4642 in Combination With Chemotherapy Versus Placebo in Combination With Chemotherapy as First-Line Therapy in Patients With Advanced or Metastatic Pancreatic Carcinoma Harboring KRAS G12D Gene Mutation
Brief Title: HRS 4642 Injection Combined With AG Versus Placebo Combined With AG Therapy in First-Line Advanced or Metastatic Pancreatic Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-4642-302
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: KRAS G12D-Mutant Advanced or Metastatic Pancreatic Cancer in the First-line Setting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRS-4642 + AG (Experimental)
  Interventions: Drug: HRS-4642 + AG
- HRS-4642 placebo + AG (Active Comparator)
  Interventions: Drug: HRS-4642 placebo + AG

INTERVENTIONS:
Drug: HRS-4642 + AG — HRS-4642 + AG
  Arms: HRS-4642 + AG
Drug: HRS-4642 placebo + AG — HRS-4642 placebo + AG
  Arms: HRS-4642 placebo + AG

SUMMARY:
This study investigates the first-line treatment of advanced pancreatic cancer with KRAS G12D mutation. Patients were randomized 1:1 to receive either the experimental regimen HRS-4642 plus AG or the control regimen AG alone.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent
2. Age 18-75 years old (inclusive) at the time of signing the informed consent form
3. Male or female
4. ECOG score of 0 or 1
5. Expected survival ≥ 12 weeks
6. At least one measurable lesion according to RECIST v1.1 criteria

Exclusion Criteria:

1. Any other condition that, in the judgment of the investigator, may increase the risk of participating in the study, interfere with the results of the study, or be unsuitable for participation in this study
2. Presence of uncontrollable psychiatric illness and other conditions such as known alcoholism, drug or substance abuse, criminal detention, etc., that affect the completion of the study procedures
3. Known hypersensitivity to any component of HRS-4642; History of severe allergic reactions to other monoclonal antibodies/fusion protein drugs; Known history of severe hypersensitivity to antineoplastic agents in combination
4. Received other major surgery other than diagnosis or biopsy within 28 days before the first dose; Minor traumatic surgery (biopsy, laparoscopy, and drainage) within 7 days prior to the first dose; Presence of non-healing wounds (severe, non-healing, or dehiscence), untreated fractures
5. Subjects who are participating in other clinical studies or whose first dose is less than 4 weeks from the end of the previous clinical study (last dose), or who have 5 half-lives of this investigational drug, whichever is shorter
6. Use of a live attenuated vaccine within 28 days prior to the first dose of study medication, or anticipated need for a live attenuated vaccine during study treatment
7. Have a history of immunodeficiency, including a positive HIV test, other acquired or congenital immunodeficiency diseases, or a history of organ transplantation
8. Those who have active pulmonary tuberculosis infection within 1 year before enrollment, or those who have a history of active pulmonary tuberculosis infection more than 1 year ago but have not been formally treated
9. Active hepatitis B
10. Presence of clinically significant acute or chronic pancreatitis
11. Poorly controlled or severe cardiovascular and cerebrovascular diseases, arterior/venous thrombotic events within 6 months prior to study entry
12. Presence of gastrointestinal obstruction or presence of symptoms and signs of gastrointestinal obstruction within 6 months prior to the start of study treatment, but screening can be performed if surgical treatment has been performed and the obstruction has been completely resolved

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 588 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
PFS as assessed by BICR per RECIST 1.1 | up to 2 years
OS | up to 3 years

SECONDARY OUTCOMES:
ORR,as assessed by BICR per RECIST v1.1 | up to 2 years
DCR as assessed by BICR per RECIST v1.1 | up to 2 years
DoR as assessed by BICR per RECIST v1.1 | up to 2 years
PFS as assessed by the investigator per RECIST v1.1. | up to 2 years
ORRas assessed by the investigator per RECIST v1.1. | up to 2 years
DCR as assessed by the investigator per RECIST v1.1. | up to 2 years
DoR as assessed by the investigator per RECIST v1.1. | up to 2 years
Incidence and severity of adverse events (AEs) graded by NCI-CTCAE v5.0. | Twice a month，up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided